CLINICAL TRIAL: NCT02926157
Title: Buying Time: Improving Sleep to Promote Cognitive Function in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H16-01029
Record Dates: First submitted 2016-09-21; First posted 2016-10-06 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Sleep; Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Life Style and Sleep Group (Experimental): Participants randomized into this group will undergo a 4 week sleep hygiene course (classes 1x/week for 1.5 hours), followed by a 20 week lifestyle activation program. During the 20 week lifestyle activation program, participants wear a Fit Bit and receive a call from a fitness professional every other week for motivation and recommendations, and receive a bright light therapy program from a sleep expert based on their initial sleep results at the baseline measurement session.
  Interventions: Behavioral: Life Style and Sleep Intervention
- Wait-list Control (No Intervention): Participants randomized into this group will complete all measurement sessions. After completion of the final measurement session (6 months), participants will be offered an abbreviated version of the Life Style and Sleep Group intervention including the sleep hygiene course, consultation with sleep expert to go over individual sleep patterns and be given recommendations, along with physical activity recommendations from a fitness expert.

INTERVENTIONS:
Behavioral: Life Style and Sleep Intervention
  Arms: Life Style and Sleep Group

SUMMARY:
The purpose of this study is to investigate whether a comprehensive group education combined with a lifestyle "activation" program that includes (a) sleep hygiene course, (b) physical activity promotion, and (c) bright light therapy, can improve both sleep quality and cognitive function among 96 community-dwelling older adults.

DETAILED DESCRIPTION:
96 community-dwelling older adults with sleep complaints will be randomized into either a 6-month life style and sleep activation intervention program or a waitlist control group (participants in this group will be offered an abbreviated version of the program upon completion of the 6 month study). There are 3 measurement sessions to measure cognition, sleep, and physical activity at the onset of the study, the midway (3 month) point, and completion (at 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Sleep complaints
* Community-dwelling (not in a long term care facility)
* Read, write, and speak English
* Able to walk independently
* In sufficient health to participate in regular physical activity

Exclusion Criteria:

* Diagnosis of obstructive sleep apnea
* Receiving continuous positive air pressure (CPAP) treatment
* Diagnosed with dementia of any type
* At high risk for cardiac complications during physical activity or unable to self-regulate activity or understand recommended activity level
* Have a clinically important peripheral neuropathy or sever musculoskeletal or joint disease that impairs mobility

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sleep quality as measured by Motion Watch 8 at 3 and 6 months | Baseline, 3 months, and 6 months

SECONDARY OUTCOMES:
Change from baseline in cognitive function as measured by the Alzheimer's Disease Assessment Scale Cognitive Subscale Plus (ADAS-Plus) at 3 and 6 months | Baseline, 3 months, and 6 months
Change from baseline in self-reported sleep quality as measured by the Pittsburgh Sleep Quality Index at 3 and 6 months | Baseline, 3 months, and 6 months
Change from baseline in physical activity levels as measured by Motion Watch 8 at 3 and 6 months | Baseline, 3 months, and 6 months
Change from baseline in self-reported physical activity levels as measured by CHAMPS physical activity questionnaire each month | Monthly, from baseline through 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Liu-Ambrose, PhD, Principal Investigator — University of British Columbia; Glenn Landry, PhD, Principal Investigator — University of British Columbia; Linda Li, PhD, Principal Investigator — University of British Columbia; Catherine Chan, MPT, Principal Investigator — University of British Columbia; John Best, PhD, Principal Investigator — University of British Columbia; Cindy Barha, PhD, Principal Investigator — University of British Columbia; Jennifer Davis, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Balbim GM, Boa Sorte Silva NC, Falck RS, Kramer AF, Voss MW, Liu-Ambrose T. 24-hour activity cycle behaviors and gray matter volume in mild cognitive impairment. Alzheimers Dement. 2025 Jul;21(7):e70496. doi: 10.1002/alz.70496. PMID 40693459
- [Derived] Falck RS, Davis JC, Best JR, Chan PCY, Li LC, Wyrough AB, Bennett KJ, Backhouse D, Liu-Ambrose T. Effect of a Multimodal Lifestyle Intervention on Sleep and Cognitive Function in Older Adults with Probable Mild Cognitive Impairment and Poor Sleep: A Randomized Clinical Trial. J Alzheimers Dis. 2020;76(1):179-193. doi: 10.3233/JAD-200383. PMID 32444553
- [Derived] Falck RS, Davis JC, Best JR, Li LC, Chan PCY, Wyrough AB, Landry GJ, Liu-Ambrose T. Buying time: a proof-of-concept randomized controlled trial to improve sleep quality and cognitive function among older adults with mild cognitive impairment. Trials. 2018 Aug 17;19(1):445. doi: 10.1186/s13063-018-2837-7. PMID 30119694